CLINICAL TRIAL: NCT03776513
Title: Impact of Juvenile Obesity on Emotional Memory and Functional Connectivity Between the Amygdala and the Hippocampus
Brief Title: Neuro-cognitive Impact of Juvenile Obesity
Acronym: OBETEEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Equipe NeuroImagerie et Cognition Humaine CNRS UMR 5287 - INCIA (Unknown); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2017/19
Record Dates: First submitted 2018-11-07; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Pediatric Obesity; Behavior and Behavior Mechanisms; Emotions
Keywords: obesity, teenagers, emotional memory, brain networks
MeSH Terms: conditions — Pediatric Obesity; Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Thirty obese boys (12-17 years old) undergoing an MRI, a clinical and psychological examination and a series of cognitive tests
  Interventions: Behavioral: an MRI examination
- control group (Other): Thirty healthy boys (12-17 years old) paired for pubertal stage, level of education and socio-economic level undergoing an MRI, a clinical and psychological examination and a series of cognitive tests
  Interventions: Behavioral: an MRI examination

INTERVENTIONS:
Behavioral: an MRI examination — The MRI examination implies the realization of an emotional associative memory task
  Other Names: a clinical and psychological examination and a series of cognitive tests

SUMMARY:
Recent studies indicate that obese teenagers exhibit memory disturbances. Adolescence represents a crucial period in the development of the hippocampus and the amygdala, necessary for the implementation of memory and emotional functions for the rest of life. Disturbances of the interaction between amygdala and hippocampus during adolescence have been associated with the development of neuropsychiatric disorders. However, the impact of juvenile obesity on functional amygdala-hippocampus connectivity has not been evaluated yet. The main objective of this study is to compare the emotional memory performance and the level of functional connectivity between the hippocampus and the amygdala during the realization of an emotional associative memory task, in obese and control adolescents.

DETAILED DESCRIPTION:
Obesity increases the prevalence of cognitive impairment. In particular, it can promote disturbances of contextual memory dependent on the hippocampus. Obesity is also associated with negative emotional consequences. However, no clinical study has so far evaluated the effect of obesity on emotional memory, a function underpinned by the amygdala. Recent studies indicate that obese children and adolescents exhibit memory disturbances. Adolescence represents a crucial period in the development of the hippocampus and the amygdala, two brain regions implicated in memory and emotional functions for the rest of life. Changes in connectivity during development, whether structural or functional, are major before the age of 10 and progressive and minor until the age of 30. Disturbances of this amygdala-hippocampal functional connectivity during adolescence have been associated with the development of neuropsychiatric disorders. However, the impact of childhood obesity on functional amygdala-hippocampus connectivity has still not been evaluated. The first aim of the study is to compare the functional connectivity of the hippocampus and the amygdala measured during the realization of an emotional associative memory task or at rest before and after the task between obese teenagers and control teenagers and how closely it is related to emotional memory performances. Secondly, it will be determined whether the level of functional connectivity between the hippocampus and the amygdala is related to cognitive performances and eating symptomatology in obese teenagers.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group: 12-17 years old boys, BMI>30 (according to IOTF), right-handed, French secondary school, beneficiary of social security, consent of the holders of parental authority.
* Control group: 12-17 years old boys, BMI<25 (according to IOTF), right-handed, French secondary school, beneficiary of social security, consent of the holders of parental authority.

Exclusion Criteria:

* Adolescent with pubertal stage of Tanner <2
* Adolescent with known visual or auditory difficulties
* Adolescent with a known chronic pathology requiring medication
* Adolescent with psychotic, neurodevelopmental or substance use disorder
* Adolescent who may have a contraindication to the MRI examination (presence in the body of metallic prostheses, pacemaker, metal chips, claustrophobia).

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-11-12 (Estimated); Study Completion 2020-12-12 (Estimated)

PRIMARY OUTCOMES:
the level of connectivity between the amygdala and the hippocampus recorded during the execution of an emotional memory task in the scanner. | through study completion, an average of 24 months
  The level of connectivity between the hippocampus and the amygdala during the performance of the task will be measured through the fluctuations of the blood oxygen level-dependent (BOLD) signal obtained in activation functional magnetic resonance imaging (fMRI) during the performance of an associative emotional memory task. The level of functional connectivity between two brain regions will be deduced from the temporal correlation between the fluctuations of the BOLD signal between these two regions. This coefficient will be normalized in Z-score before analysis.

SECONDARY OUTCOMES:
The level of connectivity between the amygdala and the hippocampus before and after the task will also be recorded at rest. | through study completion, an average of 24 months
  The level of functional connectivity at rest will be measured before and after the task performed in the scanner. The fluctuations of the BOLD signal recorded at rest (while the subject is quietly resting eyes closed in the machine without being engaged in the performance of a task) also makes it possible to measure levels of functional connectivity of rest between two brain regions according to a method a little different from that applied to activation images (after filtering high frequencies). A Z-score reflecting the level of connectivity will be calculated before statistical analysis.
The score at the emotional memory task performed in the scanner will be collected | through study completion, an average of 24 months
  The behavioral performance associated with the completion of the task is collected in an e-Prime file and expressed as percentages of correct answers.
grey matter volumes (mm3) | through study completion, an average of 24 months
  The investigators will construct volumetric grey matter maps using Voxel-Based-Morphometry toolbox of SPM for each subject so as to conduct whole brain analysis.
cortical thicknesses (mm) | through study completion, an average of 24 months
  The investigators will use FreeSurfer Suite to evaluate cortical thickness for each subject.
The percentage of body fat | through study completion, an average of 24 months
  The percentage of body fat will be evaluated by a bio-impedancemetry scale that automatically provides a measure of body fat and lean mass.
" Paired Associates Learning Task " administrated through the CANTAB neuropsychological examination | through study completion, an average of 24 months
  Paired Associates Learning assesses visual memory and new learning. Administration time: 8 minutes Task format: Boxes are displayed on the screen and are "opened" in a randomised order. One or more of them will contain a pattern. The patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located. If the participant makes an error, the boxes are opened in sequence again to remind the participant of the locations of the patterns. Increased difficulty levels can be used to test high-functioning, healthy individuals.
  Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
the number of distinct words for the free-recall phase (" Verbal Recall/Recognition Memory Task " administrated through the CANTAB neuropsychological examination) | through study completion, an average of 24 months
  Verbal Recognition Memory assesses verbal memory and new learning. It measures the ability to encode and subsequently retrieve verbal information, with recall tapping into fronto-temporal networks and recognition assessing hippocampal areas.
  Administration time: 10 minutes Task format : The participant is shown a sequence of words on screen one by one. The participant is then tasked with recalling the words, whilst a rater marks which ones they remembered. In the next phase, the participant is presented with two words, one from the original list and one distractor and is asked to choose which one they have seen before, in a 2-force choice paradigm. The latter recognition phase is then repeated after a delay.
  One of the outcome measures is the number of distinct words for the free-recall phase
" Verbal Recall/Recognition Memory Task " administrated through the CANTAB neuropsychological examination | through study completion, an average of 24 months
  Verbal Recognition Memory assesses verbal memory and new learning. It measures the ability to encode and subsequently retrieve verbal information, with recall tapping into fronto-temporal networks and recognition assessing hippocampal areas.
  Administration time: 10 minutes Task format : The participant is shown a sequence of words on screen one by one. The participant is then tasked with recalling the words, whilst a rater marks which ones they remembered. In the next phase, the participant is presented with two words, one from the original list and one distractor and is asked to choose which one they have seen before, in a 2-force choice paradigm. The latter recognition phase is then repeated after a delay.
  The other outcome measures is the number of correct and incorrect responses for the immediate and delayed recognition parts of the test.
Percentage of correct and incorrect responses at the " Emotion Recognition Task " administrated through the CANTAB neuropsychological examination | through study completion, an average of 24 months
  The Emotion Recognition Task (ERT) measures the ability to identify six basic emotions in facial expressions along a continuum of expression magnitude.
  Administration time: 6-10 minutes Task format: Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).
  The first outcome measure for ERT is the percentages of correct and incorrect responses
Number of correct or incorrect responses at the " Emotion Recognition Task " administrated through the CANTAB neuropsychological examination | through study completion, an average of 24 months
  The Emotion Recognition Task (ERT) measures the ability to identify six basic emotions in facial expressions along a continuum of expression magnitude.
  Administration time: 6-10 minutes Task format: Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).
  The second outcome is the numbers of correct or incorrect response.
Response latencies at the " Emotion Recognition Task " administrated through the CANTAB neuropsychological examination | through study completion, an average of 24 months
  The Emotion Recognition Task (ERT) measures the ability to identify six basic emotions in facial expressions along a continuum of expression magnitude.
  Administration time: 6-10 minutes Task format: Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise).
  The last outcome is the response latencies
cognitive functioning of the adolescent | through study completion, an average of 24 months
  The cognitive functioning of the adolescent will also be evaluated by his parents through the raw scores on the 8 subscales of the BRIEF-C and on composite index (Behavioral Regulation Index and Metacognition Index), based on a set of the 8 raw scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

REFERENCES:
- [Result] Vertes PE, Bullmore ET. Annual research review: Growth connectomics--the organization and reorganization of brain networks during normal and abnormal development. J Child Psychol Psychiatry. 2015 Mar;56(3):299-320. doi: 10.1111/jcpp.12365. Epub 2014 Dec 1. PMID 25441756